CLINICAL TRIAL: NCT00664677
Title: Phase 1 Study of Terameprocol (EM-1421) a Survivin and Cyclin-Dependent Kinase-1 (Cdc2) Inhibitor, in Patients With Leukemia
Brief Title: Phase 1 Study of Terameprocol (EM-1421) in Patients With Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding constraints
Sponsor: Erimos Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-1421 #105
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Leukemias; Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Adult T Cell Leukemia (ATL); Chronic Myeloid Leukemia (CML-BP); Chronic Lymphocytic Leukemia (CLL); Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML)
Keywords: Adult; Leukemia; Terameprocol; Survivin; AML; ALL; ATL; CML; CLL; CMML; MDS
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — terameprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Terameprocol (EM-1421) (Experimental): Terameprocol (EM-1421) as a single agent given intravenously over 6 hours three times a week for two weeks followed by one week rest (two weeks on, one week off).
  Interventions: Drug: Terameprocol (EM-1421)

INTERVENTIONS:
Drug: Terameprocol (EM-1421) — Terameprocol (EM-1421) as a single agent given intravenously over 6 hours three times a week for two weeks followed by one week rest (two weeks on, one week off.
  Other Names: Terameprocol; EM-1421; meso-Tetra-o-Methyl Nordihydroguaiaretic Acid

SUMMARY:
This study is designed to determine the safety, maximum tolerated dose,dose limiting toxicity of Terameprocol(EM-1421)and determine the pharmacokinetics (clearance from the blood)of Terameprocol(EM-1421)given as intravenous infusion three times a week in patients with leukemia.

DETAILED DESCRIPTION:
The dose of Terameprocol (EM-1421) will be escalated in successive cohorts of 3 patients. Patients will be entered sequentially on each dose level. If none of the first 3 patients at a dose level experience first cycle drug related dose-limiting toxicity (DLT), new patients may be entered at the next higher dose level. If 1 of 3 patients experience first cycle DLT, up to 3 more patients are started at that same dose level. If 2 or more experience first cycle DLT, no further patients are started at that dose. The MTD is the highest dose level in which <2 patients of 6 develop a first cycle DLT. New dose levels may begin accrual only if all patients at the current dose level have been observed for a minimum of 3 weeks after the last infusion of Terameprocol (EM-1421). The recommended phase 2 dose (RP2D) will be the MTD unless significant clinical activity is seen below the MTD.

During the observation period of 3 weeks, additional accrual to a previously assessed lower dose level, with no documented DLTs, will be allowed with sponsor approval.

Patients will be treated three times a week, with at least one day in between infusions, for two weeks followed by one week of rest. The dose for new cohorts will be escalated from 1000, to 1500 and 2200 mg or de-escalated to 500 mg if 1000 mg exceeds the MTD. The principal investigator will consult with the sponsor to determine the appropriate dose level for a new patient. At the MTD, up to 10 additional patients may be accrued in that dose cohort to further define the toxicities and response of the agent. If the initial dose level exceeds the MTD, a fallback dose level of 500 mg will be implemented.

Patients are allowed to be treated with subsequent cycles of Terameprocol (EM-1421) until disease progression or until severe toxicities occur and side effects do not outweigh the benefit of study drug administration in the assessment of the treating physician.

Intrapatient dose escalation Intrapatient dose escalation by one dose level may be permitted, but only if at least 3 patients in the next higher dose level have been treated and have been followed for 21 days without experiencing DLT. Decisions for intrapatient dose escalation will be made jointly by the Study Sponsor, treating physician and Principal Investigator.

Terameprocol (EM-1421) as a single agent given intravenously over 6 hours three times a week for two weeks followed by one week rest (two weeks on, one week off)in the following dose cohorts starting with 1000 mg dose cohort.

Dose Level -1: 500 mg

Dose Level 1: 1000 mg

Dose Level 2: 1500 mg

Dose Level 3: 2200 mg

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmed relapsed or refractory leukemias for which no standard therapies are available that are expected to result in durable remissions. Eligible are patients with:

   * acute myeloid leukemia (AML) by WHO or FAB classification
   * acute lymphocytic leukemia (ALL)
   * adult T cell leukemia (ATL)
   * chronic myeloid leukemia in blast crisis (CML-BP) having failed Bcr-Abl specific kinase inhibitors (e.g. imatinib and/or dasatinib)
   * chronic lymphocytic leukemia (CLL)
   * poor-risk myelodysplastic syndrome (MDS) [by WHO >10% blasts or IPSS groups: Int-2, high]
   * chronic myelomonocytic leukemia (CMML)
2. ECOG performance status of 0-1
3. Negative pregnancy test within 7 days of start of study drug NOTE: Men and women of child-producing potential must use effective contraceptive methods during the study (e.g. abstinence, intrauterine device [IUD], oral contraceptive or double barrier device)
4. Written informed consent
5. In the absence of rapidly progressing disease, the interval from prior therapies to time of study drug administration should be a minimum of 3 weeks for cytotoxic agents or at least 5 half-lives for noncytotoxic agents. Persistent chronic toxicities from prior chemotherapy must not be greater than grade 1
6. Age greater than or equal to 18 years
7. Patients must have the following clinical laboratory values:

   * Serum creatinine less than or equal to 2.0 mg/dl or creatinine clearance greater than 50ml/hr
   * Total bilirubin less than or equal to 1.5x the upper limit of normal unless considered due to Gilbert's syndrome
   * Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) less than or equal to 3x the upper limit of normal unless considered due to organ leukemic involvement

Exclusion Criteria:

Patients with any one of the following criteria will not be eligible for study participation:

1. Uncontrolled intercurrent illness including, but not limited to,

   * uncontrolled infection,
   * myocardial infarction within previous 3 months,
   * symptomatic congestive heart failure (New York Heart Association Class III, IV),
   * symptomatic coronary artery disease
   * cardiac arrhythmia not controlled by medication NOTE: Patients with controlled infection on antibiotic or antifungal therapy are eligible
2. Psychiatric illness/social situations that would limit compliance with study requirements or unwillingness or inability to comply with procedures required in this protocol
3. Patients receiving any other standard or investigational treatment for their leukemia NOTE: Hydroxyurea is allowed prior to study drug start and for the first 7 days of therapy
4. Pregnant and nursing patients are excluded. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
5. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1
6. Patients with known CNS disease
7. History of allergic reactions attributed to compounds of similar chemical or biological composition to Terameprocol (EM-1421) or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety, maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of Terameprocol (EM-1421) given as intravenous infusion three times a week in patients with leukemia | Adverse events and toxicity will be assessed prior to each cycle of treatment and at times when clinically indicated.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of Terameprocol (EM-1421) given as intravenous infusion three times a week in patients with leukemia | Pharmacokinetics samples will be collected only on the first cycle of treatment with study drug from immediately prior to first study drug infusion to the end of day 12 of infusion.
To access anti-tumor activity | Pharmacodynamic (molecular markers) samples will be collected immediately prior to, day 5 pre-dose and post-dose day 12 of each cycle of study drug administration, at remission and at relapse/or end of study (whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Neil Frazer, MB, ChB, Study Director — Erimos Pharmaceutical
Locations (1):
- UNC, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to pubmed abstract of publication Tibes et al., Investigational New Drugs April 2015, Volume 33, Issue 2, pp 389-396 — http://www.ncbi.nlm.nih.gov/pubmed/25523151